CLINICAL TRIAL: NCT04628494
Title: A Randomized, Open-Label, Phase 3 Trial of Epcoritamab vs Investigator's Choice Chemotherapy in Relapsed/Refractory Diffuse Large B-cell Lymphoma (R/R DLBCL)
Brief Title: A Phase 3 Trial of Epcoritamab vs Investigator's Choice Chemotherapy in Relapsed/Refractory (R/R) Diffuse Large B-cell Lymphoma (DLBCL)
Acronym: EPCORE DLBCL-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT3013-05; 2023-504830-23-00 (EU CTIS Number); 2020-003016-27 (EudraCT Number); jRCT2021220017 (Registry Identifier: Japan Registry for Clinical Trials (jRCT)); CTR20221558 (Registry Identifier: ChinaDrugTrials.org.cn); MOH_2021-01-18_009672 (Registry Identifier: Clinical Research Site - mytrial); NL75079.056.20 (Registry Identifier: CCMO (the Netherlands)); 286972 (Other: IRAS ID; UK Research Summaries Database)
Expanded Access: NCT05733650 (Approved for marketing)
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: double-hit DLBCL; triple-hit DLBCL; follicular grade 3B; transformed DLBCL; T-cell histiocytes-rich large B cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epcoritamab (GEN3013; DuoBody®CD3xCD20) (Experimental): Epcoritamab will be administered in Cycles of 28 days until any of the discontinuation criteria is met
  Interventions: Biological: Epcoritamab
- Investigator's choice of chemotherapy (Active Comparator): R-GemOx will be administrated in Cycles of 28 days until maximum cycles completion or any of the discontinuation criteria is met
  BR will be administrated in Cycles of 21 days until maximum cycles completion or any of the discontinuation criteria is met
  Interventions: Drug: Investigator's Choice Chemotherapy

INTERVENTIONS:
Biological: Epcoritamab — Following mandatory pre-medication, participants will be administered epcoritamab as a subcutaneous injection.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Epcoritamab (GEN3013; DuoBody®CD3xCD20)
Drug: Investigator's Choice Chemotherapy — Following mandatory pre-medication, participants will be administered intravenously either BR or R-GemOx.
  Other Names: BR or R-GemOx
  Arms: Investigator's choice of chemotherapy

SUMMARY:
The purpose of this trial is to find out if epcoritamab, also known as EPKINLY™ and GEN3013, is safe and works well as treatment for participants with DLBCL that are not responding to treatment, have grown in size, or have come back following treatment with at least 1 prior systemic cancer therapy. All participants in this trial will be randomly assigned to receive either epcoritamab or a pre-specified investigator's choice (standard of care) chemotherapy (either rituximab + gemcitabine + oxaliplatin [R-GemOx], or bendamustine + rituximab [BR]). Participants must have failed or be ineligible to receive an autologous stem cell transplant (ASCT).

Epcoritamab will be injected under the skin. Investigator's choice chemotherapy will be given intravenously.

Trial details include:

* The trial duration will be up to 5 years after last participant is randomized.
* All trial participants have a 21-day screening period, a treatment period, and a follow-up period that continues until death.
* The estimated trial duration for an individual participant depends upon the treatment arm assigned:

  * Participants who receive epcoritamab will have 28-day treatment cycles. Epcoritamab will be given once weekly for the first 3 months, then every other week for 6 months, then every 28 days until lymphoma progression or unacceptable adverse events.
  * Participants who receive investigator's choice (standard of care) chemotherapy will receive treatments either:

    * R-GemOx: On Day 1 (or Day 1 & Day 2), and Day 15 (or Day 15 & Day 16) every 28 days, for up to 4 months; or
    * BR: On Day 1 and Day 2 every 3 weeks for up to 4.5 months.

DETAILED DESCRIPTION:
The trial is an open label, multi-center, global phase-3 randomized trial of epcoritamab. The goal of this randomized trial is to evaluate the efficacy of epcoritamab (GEN3013, DuoBody®-CD3xCD20) compared to investigator's choice of chemotherapy, in participants with relapsed, refractory DLBCL who have failed or are ineligible for high-dose chemotherapy and autologous stem cell transplant (HDT-ASCT). No change in chemotherapy is permitted for participants during the treatment phase of the trial.

Overall Survival (OS) is the primary endpoint in USA and in China, with the analysis population including all randomized participants. OS/Progression Free Survival (PFS) are dual-primary endpoints for rest of the world (outside US and China), with the analysis population also including all participants randomized.

The China sub-study of GCT3013-05 is registered under NCT07226752.

ELIGIBILITY:
Main Inclusion Criteria:

1. Relapsed or refractory disease and previously treated with at least 1 line of systemic antineoplastic therapy including anti-CD20 monoclonal antibody (mAb)-containing combination chemotherapy since lymphoma diagnosis
2. One of the confirmed histologies below with CD20-positivity:

   1. DLBCL, not otherwise specified (NOS), including de novo or histologically transformed from follicular lymphoma (FL)
   2. "Double-hit" or "triple-hit" DLBCL (technically classified in World Health Organization (WHO) 2016 as high-grade B-cell lymphoma (HGBCL), with MYC and BCL2 and/or BCL6 translocations), including de novo or histologically transformed from FL
   3. FL Grade 3B
   4. T-cell/histiocyte-rich large B-cell lymphoma
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-2
4. Failed previous HDT-ASCT or not eligible for high-dose therapy autologous stem cell transplant (HDT-ASCT) at screening
5. Participants must have detectable disease by positron emission tomography (PET) scan and measurable by computed tomography (CT) scan or magnetic resonance imaging (MRI)
6. Acceptable renal and liver function
7. Life expectancy >2 months on standard of care treatment

Main Exclusion Criteria:

1. Primary Central Nervous System (CNS) tumor or known CNS involvement
2. Any prior therapy with a bispecific antibody targeting CD3 and CD20
3. Major surgery within 4 weeks prior to randomization
4. Chemotherapy and other non-investigational antineoplastic agents (except CD20 mAbs) within 4 weeks or 5 half-lives (whichever is shorter) prior to randomization
5. Any investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to randomization
6. Autologous stem cell transplant (ASCT) within 100 days of randomization
7. Treatment with chimeric antigen receptor T-cell (CAR-T) therapy within 100 days prior to randomization
8. Seizure disorder requiring anti-epileptic therapy
9. Clinically significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 5 years
Overall Response Rate (ORR) | Up to approximately 5 years
Complete Response (CR) Rate | Up to approximately 5 years
Duration of Response (DOR) | Up to approximately 5 years
Time to Response (TTR) | Up to approximately 5 years
Duration of Minimal Residual Disease (MRD) Negative Status | Up to approximately 5 years
Rate of MRD Negative Status | Up to approximately 5 years
Time to Next Anti-lymphoma Therapy (TTNT) | Up to approximately 5 years
Number of Participants with Adverse Events (AEs) | Up to approximately 5 years
Number of Participants with Dose Interruptions and Delays | Up to approximately 5 years
Number of Participants with an Anti-epcoritamab Antibody Response | Up to approximately 5 years
Changes from Baseline in Lymphoma Symptoms as Measured by the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) | Baseline up to approximately 5 years

CONTACTS AND LOCATIONS:
Locations (186):
- United States (15):
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Community Health Network Cancer Center North, Indianapolis, Indiana
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Henry Ford Health System, Jackson, Michigan
  - MMCORC Attn Delaney Anderson, Saint Louis Park, Minnesota
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - TriHealth Cancer Institute- Good Samaritan Hospital, Cincinnati, Ohio
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University (VCU) Massey Cancer Center, Richmond, Virginia
  - North Star Lodge Cancer Center, Yakima, Washington
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Australia (6):
  - Flinders Medical Centre, Bedford Park
  - Concord Repatriation General Hospital, Concord
  - Peninsula Private Hospital Clinical Trials Unit, Frankston
  - Icon Cancer Centre Corporate Office, South Brisbane
  - Calvary Mater Newcastle, Waratah
  - Westmead Hospital, Westmead
- Austria (3):
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Uniklinikum Salzburg, Universitätsklinik für Innere Medizin III der PMU, Salzburg
- Belgium (9):
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Brussel, Jette
  - Hôpital de Jolimont, La Louvière
  - Universitair Ziekenhuis gasthuisberg Leuven, Leuven
  - AZ Nikolaas- Verenigde Ziekenhuizen van Waas en Durme, Sint-Niklaas
  - AZ Turnhout, Campus Sint-Elisabeth, Turnhout
- CHU de Quebec-Universite Laval, Québec, Canada
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus University Hospital, Department of Hematology, Clinical Research Unit C116, Aarhus
  - Clinical Research Unit, Roskilde Sygehus, Roskilde
  - Vejle Hospital, Vejle
- Finland (2):
  - HUS Cancer Center/ Clinical Trial Unit, Helsinki
  - Oulu university hospital, Department of hematology, Oulu
- France (19):
  - Audrey ALEME, Amiens
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHRU de Brest - Hospital Morvan, Brest
  - CHU Caen - IHBN, Caen
  - Groupe Hospitalier de La Rochelle, La Rochelle
  - CHU de LIMOGES, Limoges
  - Centre Léon Bérard, Lyon
  - Hopital de la Conception APHM, Marseille
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Clinique Victor Hugo, Paris
  - Hôpital Saint-Louis, Paris
  - CHU de Bordeaux Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital la Milétrie, Poitiers
  - Centre Hospitalier Rene Dubos, Pontoise
  - Ch Cornouaille, Quimper
  - Centre Henri Becquerel, Rouen
  - CHRU Tours Hôpital Bretonneau, Tours
- Germany (4):
  - Uniklinik Köln, Klinik I für Innere Medizin, CIO Gebäude 70, 5.094, Cologne
  - Universitaetsklinikum Essen, Essen
  - Universitätsklinikum Schleswig-Holstein Medizinische Klinik II Hämatologie und Onkologie, Kiel
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (9):
  - National Institute of Oncology, Budapest
  - Semmelweis Egyetem Belgyógyászati és Onkológiai Klinika, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Belgyogyaszati Klinika, Hematologia, Debrecen
  - Belgyógyászati osztály Markhot Ferenc Kórház, Eger
  - Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Josa Andras Teaching Hospital, Hematology Dept, Nyíregyháza
  - University of Pecs 1st. Internal medicine Clinic Dept. Hematology, Pécs
  - Szegedi Tudományegyetem II. sz. Belgyogyaszat, Hematologia, Szeged
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Italy (13):
  - IRCCS Istituto Tumori Giovanni Paolo II Bari, Bari
  - Azienda Socio Sanitaria Territoriale Sette Laghi (Presidio Ospedale di Circolo e Fondazione Macchi), Bergamo
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola
  - Istituto Oncologico Europeo, Milan
  - San Raffaele Hospital, Milan
  - Azienda Ospedaliero - Universitaria Maggiore delle Carita SCDU Ematologia building C, Novara
  - Fondazione IRCCS Policlinico San matteo, Pavia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Azienda Ospedaliera Universitaria Policlinico Umberto I Università di Roma La Sapienza, Dip Med Tra, Rome
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI) Ospedale Maggiore di Trieste, Trieste
  - SC di Ematologia - AON SS Antonio e Biagio e Cesare Arrigo, Venezia
- Japan (18):
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Chugoku Central Hospital, Fukuyama
  - Hokkaido University Hospital, Hokkaido
  - National Cancer Center Hospital East, Kashiwa
  - Kyoto University Medical Hospital, Kyoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - Mie University Hospital, Mie
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - NHO Nagoya Medical Center, Nagoya
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Ōsaka-sayama
  - Tohoku University Hospital, Sendai
  - Keio University Hospital, Tokyo
  - National Cancer Center Hospital, Tokyo
  - Tokai University Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - Yamagata University Hospital, Yamagata
- Netherlands (7):
  - Rijnstate Arnhem, Arnhem
  - Amphia Ziekenhuis, Interne Geneeskunde, Oncologie. Route 43, Breda
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Bravis Ziekenhuis, Roosendaal
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis And Vlietland, Rotterdam
- Norway (2):
  - Oslo University Hospital location Radium hospital, Oslo
  - St. Olavs Hospital HF, Trondheim
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Kraków, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii, Lodz
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Russia (6):
  - State Autonomous Institution of Healthcare Republican Clinical Oncological Dispensary of the Ministr, Kazan'
  - Federal State Budgetary Institution of Science, Moscow
  - Federal State Budgetary Institution, Moscow
  - State Budgetary Institution of Healthcare of Nizhniy Novgorod region, 1st inpatient facility, 5th fl, Nizhny Novgorod
  - Federal State Budgetary Institution V.A. Almazov National Medical Research Center of the Ministry of, Saint Petersburg
  - State Budgetary Institution of Healthcare Leningrad Regional Clinical Hospital, Saint Petersburg
- Singapore (3):
  - National University Hospital, Kent Ridge
  - Clinical Trials and Research Centre, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (12):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Pusan National University Hosptial, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Chonbuk National University Hospital, Geumam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St. Marys Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (15):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospita Universitario Puerta Del Mar, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Md Anderson Cancer Center, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen De Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
- Karolinska university Hospital, Stockholm, Sweden
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (11):
  - Ankara University Medical Faculty, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Gazi University Medical Faculty, Ankara
  - Amerikan Hospital, Istanbul
  - Iqvia Tibbi Istatistik, Istanbul
  - Istanbul University Cerrahpasa - Cerrahpasa Tip Fakultesi, Istanbul
  - Istanbul University Medical Faculty, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Ege University Medical Faculty, Izmir
  - Tekirdag Namik Kemal University, Tekirdağ
  - Karadeniz Technical University, Trabzon
- United Kingdom (9):
  - Haematology - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Guys and St Thomas NHS Foundation Trust, London
  - Hammersmith Hospital, London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital, Plymouth
  - University Hospital Southampton, Southampton
  - Royal Marsden NHS Foundation Trust (Sutton), Sutton
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No